CLINICAL TRIAL: NCT03425981
Title: EFFECTS OF WHOLE-BODY ELECTROMYOSTIMULATION TRAINING ON HEALTH AND PERFORMANCE PARAMETERS IN RECREATIONAL RUNNERS.
Brief Title: Effects of WB-EMS in Runners.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Manuel Castillo Garzón, University professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 200/CEIH/2016
Record Dates: First submitted 2018-01-26; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Physical Activity
Keywords: WB-EMS; Running economy; VO2max
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WB-EMS-SRT (Experimental): Training with basic global electrostimulation
  Interventions: Other: Whole-Body Electromyostimulation Training
- WB-EMS-WT (Experimental): Training with specific global electrostimulation for runners
  Interventions: Other: Whole-Body Electromyostimulation Training
- CG (Placebo Comparator): The participants in the control group will maintain the volume and intensity of the training prior to the intervention study and the subjects of the WB-EMS and WB-EMS-AC groups will substitute one conventional training day for one with global electrostimulation for six weeks; the training of the first group will be non-specific and that of the second specific for runners and the duration of both will be 20 minutes.
  Interventions: Other: Whole-Body Electromyostimulation Training

INTERVENTIONS:
Other: Whole-Body Electromyostimulation Training — The WB-EMS training program consisted of six WB-EMS training sessions (one per week) and six running training sessions (also one per week).
  This intervention programme followed a within-day undulating periodization model. The training sessions were divided into four parts: warm up (A), strength (B), high intensity interval power training (c), and high intensity interval training (HIIT) (D).

SUMMARY:
The subjects will be randomly distributed into 3 experimental groups: training with basic global electrostimulation (WB-EMS-SRT), training with specific global electrostimulation for runners (WB-EMS-WT) and control group (CG).

Initially and at the end of the intervention period, which will consist of six weeks, the subjects will undergo a series of tests: (1) Maximum incremental effort test in tapestry to exhaustion to determine cardiorespiratory capacity (VO2max) and thresholds (aerobic and anaerobic). (2) Submaximal carpet test at constant speed to determine race economy (EC). (3) Lower train power test (CMJ and Abalakov). (4) Weight, size and waist circumference. The aforementioned tests will be carried out on different days to avoid the effect of fatigue on performance with a break of more than 48 hours between tests.

The participants in the control group will maintain the volume and intensity of the training prior to the intervention study and the subjects of the WB-EMS and WB-EMS-AC groups will substitute one conventional training day for one with global electrostimulation for six weeks; the training of the first group will be non-specific and that of the second specific for runners and the duration of both will be 20 minutes.

DETAILED DESCRIPTION:
A randomized controlled trial design was applied following CONSORT statements. After baseline measurements, participants were randomized into two groups: (i) WB-EMS group and (ii) Control Group (CG). Participants in the WB-EMS group were instructed to reduce their running training program volume, whereas the CG continued with their running training in term of volume and intensity: two or three times per week (45-60 minutes per day) at an intensity of 60-70% hearth rate reserve, which was controlled by heart rate monitor (Polar RS300X, POLAR, Kempele, Finland), and with 24-48 hours of rest between sessions

ELIGIBILITY:
Inclusion Criteria:

* Frequent runners

Exclusion Criteria:

* Received WB-EMS training.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen consumption | Baseline and through study completion, an average of 5 weeks
  Maximal Oxygen consumption was assessed using a maximum treadmill (H/P/ Cosmos Pulsar treadmill, H/P/Cosmos Sport & Medical GMBH, Germany) exercise test with a progressive incremental protocol that has been used.

SECONDARY OUTCOMES:
Ventilatory thresholds | Baseline and through study completion, an average of 5 weeks
  VT1 and VT2 were estimated from gas exchange data through different respiratory variables: minute ventilation (VE) and equivalents for oxygen (VE/VO2) and carbon dioxide (VE/VCO2) by two independent researchers
Running economy | Baseline and through study completion, an average of 5 weeks
  RE was determined during a treadmill test following a specific protocol used in previous studies
Muscular power | Baseline and through study completion, an average of 5 weeks
  Vertical jump performance was assessed using the Bosco Test.
Weight | Baseline and through study completion, an average of 5 weeks
  Weight in Kilograms
Body composition | Baseline and through study completion, an average of 5 weeks
  Assessed using DXA.

CONTACTS AND LOCATIONS:
Overall Officials: Baseline and post Castillo Garzón, University Proffesor, Study Director — Universidad de Granada
Locations (1):
- Medicine Faculty, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided